CLINICAL TRIAL: NCT04667949
Title: A 24-month, Open-label, Prospective, Multicenter Interventional, Single-arm Study Assessing the Efficacy and Safety of Fingolimod (Gilenya) 0.5 mg in Relapsing Multiple Sclerosis (RMS) Patients in China
Brief Title: Study of Efficacy and Safety of Fingolimod (Gilenya) 0.5 mg in Chinese Patients With Relapsing Multiple Sclerosis (RMS) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720D2419; 2024-000601-32 (EudraCT Number)
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
Keywords: Relapsing Multiple Sclerosis (RMS); Fingolimod; Adult; Pediatric; China
MeSH Terms: interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fingolimod (Experimental): Fingolimod 0.5 mg capsule taken orally once daily
  Interventions: Drug: Fingolimod 0.5mg

INTERVENTIONS:
Drug: Fingolimod 0.5mg — Subjects received fingolimod 0.5mg capsule QD up to month 24
  Other Names: FTY720

SUMMARY:
The main purpose of this study was to assess the efficacy and safety of 0.5mg Fingolimod (Gilenya) in Chinese patients with relapsing multiple sclerosis (RMS)

DETAILED DESCRIPTION:
This was a 24-month, open-label, multicenter, interventional, single-arm study to collect efficacy and, safety of oral fingolimod 0.5 mg/day in approximately 100 relapsing multiple sclerosis (RMS) participants in China.

The study consisted of three Phases:

* Screening (up to 1 month): After signing informed consent, participants entered a Screening Phase to determine eligibility according to inclusion and exclusion criteria.
* Treatment Period (24 months): On visit Day 1, all eligibility criteria were confirmed, including a pre-dose ECG and vital signs. The first dose of study drug was taken in the clinic on Day 1 and the participant was monitored for 6 hours after the first dose administration before discharge. Participants returned to site for evaluation at month 1 and then every three months until the end of treatment up to 24 months.
* Follow Up (2 months): Subjects who completed Treatment Period or discontinued from treatment returned for the Follow-up visit 2 months after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participant 10 to 17 years old inclusive with weight > 40kg.
* Participant 18 to 65 years old inclusive;
* Participants with relapsing multiple sclerosis
* Participants never used fingolimod before enrollment
* Subjects with Expanded Disability Status Scale (EDSS) score of 0 - 6.0 (inclusive) at Screening

Exclusion Criteria:

* Participants with certain cardiovascular conditions and/or findings in the screening ECG.
* Diagnosis of macular edema during screening visit.
* Increased risk for opportunistic infections
* Participants with known active malignancies.
* Participants who have been treated with teriflunomide within 3.5 months prior to baseline, except if active washout.
* Participants with severe active infections, active chronic infection.
* Participants with severe liver impairment.
* Pregnant confirmed by a positive pregnancy test or nursing (lactating) women.

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 13 sites in China
Pre-assignment Details: There were up to 30 days of screening period (day -30 to -1) before first treatment (day 1).
Groups:
- Fingolimod (< 18 Years): Fingolimod 0.5 mg capsule taken orally once daily in participants under 18 years old
- Fingolimod > 18 Years: Fingolimod 0.5 mg capsule taken orally once daily in participants 18 years old or over
Period: Overall Study
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Started | 11 | 87
Completed | 10 | 75
Not Completed | 1 | 12
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Subject decision | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years | Total
Number analyzed (Participants) | 11 | 87 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (1.60) | 32.3 (9.11) | 30.1 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 51 | 54
  Male | 8 | 36 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 87 | 98
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Age categorical [Count of Participants; unit: Participants]
  Children 2-11 years | 2 | 0 | 2
  Adolescents 12-17 years | 9 | 0 | 9
  Adults 18-64 years | 0 | 87 | 87
Number of relapses in the last 12 months prior to screening [Mean (Standard Deviation); unit: relapses/year] | 1.7 (1.27) | 1.2 (0.47) | 1.3 (0.62)
Number of relapses in 12 to 24 months prior to screening [Mean (Standard Deviation); unit: relapses/year] | 0.8 (1.25) | 0.7 (0.84) | 0.7 (0.89)

OUTCOME MEASURES:

1. Post Hoc Outcome: Participant Based Annualized Relapse Rate (ARR)
Description: A relapse is an appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event which is present for at least 24 hours in the absence of fever or infection.
  A relapse is confirmed by the treating physician when it is accompanied by an increase of at least 0.5 on the Expanded Disability Status Scale (EDSS) or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS).
  Participant-based ARR was calculated by taking the total number of relapses observed for a participant divided by the total number of days in study of that participant and multiplied by 365.25.
Time Frame: Baseline to Month 24
Population: Full Analysis Set (FAS): all participants who had signed the Informed Consent and who had received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: relapses per participant-year
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 11 | 87
relapses per participant-year
  All relapses - Participant based | 0.1952 (0.50314) | 0.0969 (0.50002)
  Confirmed relapses - Participant based | 0.0460 (0.15253) | 0.0372 (0.24424)

2. Post Hoc Outcome: Time Based Annualized Relapse Rate (ARR)
Description: A relapse is an appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event which is present for at least 24 hours in the absence of fever or infection. A relapse is confirmed by the treating physician when it is accompanied by an increase of at least 0.5 on the Expanded Disability Status Scale (EDSS) or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS).
  Time-based ARR was calculated by taking the total number of relapses observed for all subjects within an age group divided by the total number of days in study of all subjects within the group and multiplied by 365.25 days.
Time Frame: Baseline to Month 24
Population: as for outcome 1
Measure: Number; unit: relapses per participant-year
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 11 | 87
relapses per participant-year
  All relapses - Time based | 0.161 | 0.065
  Confirmed relapses - Time based | 0.054 | 0.019

3. Primary Outcome: Adjusted Annualized Relapse Rate (ARR) in Adult Group
Description: A confirmed relapse is any relapse that is accompanied by an increase of at least 0.5 on the EDSS or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS) as confirmed by the treating physician.
  The adjusted annualized relapse rate (ARR) was estimated by a negative binomial regression model with log-link function, the cumulative number of confirmed MS relapses per subject as the response variable, number of relapses in the previous two years before enrollment and baseline EDSS as continuous covariates. Natural log of time on study in years was used as the offset variable to account for the varying lengths of subjects' time in the study. The adjusted ARR (i.e.model-based estimate adjusted for covariates) and the corresponding 95% confidence interval were obtained.
  As per SAP this analysis was only performed for the Adult group. Descriptive data is presented in subsequent OMs.
Time Frame: Baseline to Month 24
Population: Adult participants in the Full Analysis Set (FAS). FAS: all participants who had signed the Informed Consent and who had received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Fingolimod > 18 Years
Number analyzed (Participants) | 87
relapses per participant-year | 0.018 [0.006 to 0.061]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject after providing written informed consent for participation in the study.
  For reporting purposes, the main focus was on treatment emergent adverse event (TEAE), defined as any AE which started on or after the day of first dose of study medication or events present prior to the start of treatment but increased in severity.
Time Frame: From first dose of study treatment to 45 days after last study dose up to aproximately 25.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 11 | 87
Participants
  Adverse events (AEs) | 11 | 86
  Study treatment related AEs | 10 | 81
  Serious adverse events (SAEs) | 3 | 12
  AEs leading to interruption of study treatment | 3 | 11
  AEs leading to study discontinuation | 1 | 5
  AEs leading to death | 0 | 0

5. Secondary Outcome: Annualized Rate of the Number of New or Newly Enlarged T2 Lesions
Description: Obtained from fitting a negative binomial regression model with log-link function, the total number of new or newly enlarged T2 lesions during the treatment period (per participant) as the response variable.
  The model included baseline age and volume of T2 lesions at baseline as continuous covariates. Natural log of time from screening scan in years was used as the offset.
  Baseline is defined as the last non-missing assessment obtained prior to the first administration of study drug. As per SAP this analysis was only performed for the Adult group.
Time Frame: Baseline to end of treatment (up to Month 24)
Population: Adult participants in the Full Analysis Set (FAS) with available data for the outcome measure.. FAS: all participants who had signed the Informed Consent and who had received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Lesions per participant-year
Arm/Group | Fingolimod > 18 Years
Number analyzed (Participants) | 81
Lesions per participant-year | 1.316 [0.762 to 2.272]

6. Secondary Outcome: Change From Baseline in Number of New or Newly Enlarged T2 Lesions
Description: Number of new/newly enlarged T2 lesions since baseline as measured by MRI
Time Frame: Baseline up to Month 24
Population: Participants in the Full Analysis Set (FAS) with available data for the outcome measure. FAS: all participants who had signed the Informed Consent and who had received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: new / newly enlarged T2 lesions
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 10 | 81
new / newly enlarged T2 lesions
  12 months: number analyzed (Participants) | 10 | 79
  12 months | 1.8 (1.93) | 1.8 (4.18)
  24 months | 2.1 (2.18) | 2.4 (4.84)

7. Secondary Outcome: Change From Baseline in T2 Lesion Volume
Description: T2 lesion volume as measured by MRI and calculated as post-baseline value - baseline value
Time Frame: Baseline up to Month 24
Population: Participants in the Full Analysis Set (FAS) with non-missing, non-zero baseline and post-baseline values for the outcome measure. FAS: all participants who had signed the Informed Consent and who had received at least one dose of study treatment.
Measure: Median (Full Range); unit: milliliters
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 10 | 79
milliliters
  12 months | 0.6140 [-17.607 to 34.748] | 0.3930 [-6.343 to 25.158]
  24 months: number analyzed (Participants) | 8 | 73
  24 months | -1.6736 [-17.100 to 36.719] | 0.4065 [-5.741 to 26.322]

8. Secondary Outcome: Number of Gd-enhancing T1 Lesions Per Scan in Adult Group
Description: Obtained from fitting a negative binomial regression model with log-link function, the total number of Gd-enhancing T1 lesions during the treatment period (per patient) as the response variable.
  The model included baseline age and number of Gd-enhancing T1 lesions at baseline as continuous covariates. Natural log of the number of MRI scans was used as the offset.
  MRI scans were performed at baseline, month 12 and month 24 and End of treatment for participants that discontinued treatment. Unscheduled MRIs could be performed at the investigator's judgement. As per SAP this analysis was only performed for the Adult group.
Time Frame: Baseline up to Month 24
Population: Adult participants in the Full Analysis Set (FAS) with available data for the outcome measure. FAS: all participants who had signed the Informed Consent and who had received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Lesions per participant per scan
Arm/Group | Fingolimod > 18 Years
Number analyzed (Participants) | 80
Lesions per participant per scan | 0.376 [0.216 to 0.655]

9. Secondary Outcome: Number of Gd-enhancing T1 Lesions
Description: Number of Gd-enhancing T1 lesions as measured by MRI
Time Frame: Baseline up to Month 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T1 lesions
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 10 | 79
T1 lesions
  12 months | 0.4 (0.70) | 0.4 (0.84)
  24 months: number analyzed (Participants) | 8 | 73
  24 months | 0 (0.00) | 0.4 (1.83)

10. Secondary Outcome: Change From Baseline in Gd-enhancing T1 Lesion Volume
Description: Gd-enhancing T1 lesion volume as measured by MRI and calculated as post-baseline value - baseline value
Time Frame: Baseline up to Month 24
Population: as for outcome 7
Measure: Median (Full Range); unit: microliters
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 10 | 79
microliters
  12 months | -56.0 [-1392.5 to 418.0] | 0.00 [-1869.0 to 546.0]
  24 months: number analyzed (Participants) | 8 | 73
  24 months | -56.0 [-632.7 to 0.0] | 0.00 [-1869.0 to 1082.0]

11. Secondary Outcome: Number of T1 Hypo-intense Lesions
Description: Number of T1 hypo-intense lesions as measured by MRI
Time Frame: Baseline up to Month 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T1 hypo-intense lesions
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 10 | 79
T1 hypo-intense lesions
  12 months | 14.6 (12.97) | 17.0 (13.62)
  24 months: number analyzed (Participants) | 8 | 73
  24 months | 13.4 (10.86) | 16.7 (13.27)

12. Secondary Outcome: Change From Baseline in T1 Hypo-intense Lesion Volume
Description: T1 hypo-intense lesions as measured by MRI and calculated as post-baseline value - baseline value
Time Frame: Baseline up to Month 24
Population: as for outcome 7
Measure: Median (Full Range); unit: microliters
Arm/Group | Fingolimod (< 18 Years) | Fingolimod > 18 Years
Number analyzed (Participants) | 10 | 79
microliters
  12 months | -77.500 [-6849.30 to 20341.80] | 44.000 [-4921.30 to 19035.00]
  24 months: number analyzed (Participants) | 8 | 73
  24 months | -641.415 [-7444.50 to 1161.50] | 187.100 [-5772.20 to 19264.00]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment to 60 days after last study dose up to approximately 26 months
Groups:
- Less Than 18 Years: Less than 18 years
- Greater Than or Equal to 18 Years: Greater than or equal to 18 years
- Overall: Overall
Arm/Group | Less Than 18 Years | Greater Than or Equal to 18 Years | Overall
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/87 | 0/98
Serious Adverse Events (participants affected / at risk) | 3/11 | 12/87 | 15/98
Other Adverse Events (participants affected / at risk) | 11/11 | 85/87 | 96/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Less Than 18 Years (N=11) | Greater Than or Equal to 18 Years (N=87) | Overall (N=98)
Iridocyclitis (Eye disorders) | 0 | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 2 | 2
Liver injury (Hepatobiliary disorders) | 0 | 3 | 3
COVID-19 (Infections and infestations) | 0 | 2 | 2
Febrile infection (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Acute disseminated encephalomyelitis (Nervous system disorders) | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 2 | 0 | 2
Syncope (Nervous system disorders) | 1 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Less Than 18 Years (N=11) | Greater Than or Equal to 18 Years (N=87) | Overall (N=98)
Hypoglobulinaemia (Blood and lymphatic system disorders) | 1 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 5 | 22 | 27
Lymphopenia (Blood and lymphatic system disorders) | 7 | 24 | 31
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 5
Sinus bradycardia (Cardiac disorders) | 0 | 13 | 13
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1 | 2
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 1
Ocular hypertension (Eye disorders) | 1 | 0 | 1
Refraction disorder (Eye disorders) | 1 | 0 | 1
Strabismus (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 8
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Chest discomfort (General disorders and administration site conditions) | 1 | 0 | 1
Chest pain (General disorders and administration site conditions) | 1 | 2 | 3
Influenza like illness (General disorders and administration site conditions) | 1 | 3 | 4
Pyrexia (General disorders and administration site conditions) | 4 | 12 | 16
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 10 | 10
Bronchitis (Infections and infestations) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 35 | 37
Gingivitis (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 9 | 13
Pharyngitis (Infections and infestations) | 4 | 0 | 4
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 21 | 25
Urinary tract infection (Infections and infestations) | 0 | 16 | 16
Alanine aminotransferase increased (Investigations) | 2 | 33 | 35
Aspartate aminotransferase increased (Investigations) | 1 | 19 | 20
Blood cholesterol increased (Investigations) | 1 | 1 | 2
Electrocardiogram PR shortened (Investigations) | 1 | 3 | 4
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0 | 1
Electrocardiogram high voltage (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 10 | 10
Liver function test abnormal (Investigations) | 2 | 0 | 2
Lymphocyte count decreased (Investigations) | 2 | 53 | 55
Lymphocyte percentage decreased (Investigations) | 1 | 7 | 8
Monocyte count increased (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 4 | 6
Neutrophil percentage increased (Investigations) | 1 | 1 | 2
Platelet count increased (Investigations) | 1 | 2 | 3
Protein urine present (Investigations) | 2 | 1 | 3
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 1
Urinary sediment present (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 5 | 8 | 13
Weight increased (Investigations) | 4 | 8 | 12
White blood cell count decreased (Investigations) | 4 | 22 | 26
White blood cell count increased (Investigations) | 1 | 1 | 2
White blood cells urine positive (Investigations) | 2 | 8 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 9 | 9
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 5
Headache (Nervous system disorders) | 2 | 10 | 12
Seizure (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 2
Initial insomnia (Psychiatric disorders) | 1 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 1
Urine abnormality (Renal and urinary disorders) | 1 | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 6 | 6
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT04667949/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT04667949/SAP_001.pdf